CLINICAL TRIAL: NCT04302103
Title: A Study of RC18, a Recombinant Human B Lymphocyte Stimulator Receptor:Immunoglobulin G( IgG ) Fc Fusion Protein for Injection for the Treatment of Subjects With Systemic Myasthenia Gravis
Brief Title: A Study of TACI（Transmembrane Activator and Calcium-modulator and Cyclophilin Ligand (CAML) Interactor）-Antibody Fusion Protein Injection (RC18) in Subjects With Systemic Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18C011
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Systemic Myasthenia Gravis
MeSH Terms: interventions — RC-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC18 160mg (Experimental): Patients received the test group RC18 160mg weekly administered subcutaneously for 24 times.
  Interventions: Biological: RC18 160mg
- RC18 240 mg (Experimental): Patients received the test group RC18 240mg weekly administered subcutaneously for 24 times.
  Interventions: Biological: RC18 240 mg

INTERVENTIONS:
Biological: RC18 160mg — subcutaneous injection
  Arms: RC18 160mg
Biological: RC18 240 mg — subcutaneous injection
  Arms: RC18 240 mg

SUMMARY:
The purpose of this study is to initially observe the safety and effectivity of RC18 in Participants with systemic myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent ;
2. Patient diagnosed with systemic myasthenia gravis according to The following conditions.
3. Seropositive at screening for AChR（Acetylcholine receptor）-Ab or MuSK（Muscle specific tyrosine kinase）-Ab;
4. MGFA（Myasthenia Gravis Foundation of America） Clinical classification Ⅱ-IIIb;
5. QMG score≥8,and QMG score>2 in four or more items;
6. Maintained any one of the stable standard treatment programs in the trial protocol.

Exclusion Criteria:

1. Combined autoimmune diseases, such as systemic lupus erythematosus,rheumatoid arthritis, systemic sclerosis and so on,except for hypothyroidism and hyperthyroidism;
2. Abnormal laboratory parameters need to be excluded, including but not limited to:
3. Immunosuppressive agents except agents of standard treatment programs were used within one month prior to randomization.;
4. Use of biological agents for targeted therapy within 6 months prior to randomization;
5. Intravenous immunoglobulin therapy or plasma exchange therapy within 2 months before randomization;
6. Active infection during screening(For example,herpes zoster,HIV antibody positive,active tuberculosis,etc);
7. Currently suffering from active hepatitis or severe liver lesions and history;
8. Diabetics with poor blood sugar control:HbAlc>9.0% or FBG≥11.1mmol/L;
9. Currently having a thymic tumor ,or had a thymectomy within 6 months prior to screening;
10. Received live vaccines within 3 months before randomization,or scheduled to administer vaccine during the trial;
11. Malignant tumor patients;
12. Allergic to human biological preparations;
13. Have participated in any clinical trial within 28 days before randomization,or in 5 times half-life period of the drugs of any clinical trial(taking the longer time).
14. Pregnant , lactating women and men or women who have birth plans during the research;
15. Having alcohol or drug abuse that affect the experimental conditions;
16. Investigator considers candidates not appropriating for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
The average variation of QMG scores of the twenty-fourth week compared to the QMG scores of baseline | week 24
  QMG score=Quantitative Myasthenia Gravis Score

SECONDARY OUTCOMES:
The average variation of clinical absolute score for myasthenia gravis of the twelfth and twenty-fourth weeks compared to Clinical absolute score for myasthenia gravis of baseline | week 12，24
  It is best that the assessors in each center are fixed during the study.
The average variation of QMG score of the twelfth week compared to the OMG scores of baseline | week 12
  QMG score=Quantitative Myasthenia Gravis Score

CONTACTS AND LOCATIONS:
Overall Officials: Xianhao Xu, M.D., Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Tiantan Hospital,Capital Medical University, Beijing, Beijing Municipality, China